CLINICAL TRIAL: NCT03597347
Title: An Open-label, Non-controlled, Multicenter, Pilot Trial, Using Inhaled Molgramostim in Cystic Fibrosis Subjects With Nontuberculous Mycobacterial (NTM) Infection
Brief Title: Trial of Inhaled Molgramostim in Cystic Fibrosis Subjects With Nontuberculous Mycobacterial Infection
Acronym: ENCORE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment for trial stopped early due to limitations from COVID-19, additionally changes in the standard of care for CF patients during the study period resulted in confounding of the primary endpoint.
Sponsor: Savara Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAV008-02
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Results first posted 2021-10-11 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Mycobacterium Infections, Nontuberculous; Cystic Fibrosis (CF)
Keywords: Nontuberculosis mycobacterial infection; Cystic fibrosis; M. avium complex; M. abscessus complex; Mycobacterium Infections, Nontuberculous
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous; Cystic Fibrosis | interventions — regramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Group 1 (Experimental): Participants with chronic pulmonary MAC or MABSC infection who have not consistently achieved negative NTM sputum cultures while currently on a multidrug NTM guideline-based antimycobacterial regimen, which has been ongoing for at least 9 months prior to the Baseline visit.
  Interventions: Drug: Molgramostim nebulizer solution; Device: PARI eFlow nebulizer system
- Group 2 (Experimental): Participants with chronic pulmonary MAC or MABSC infection who remain sputum culture positive but have stopped a multidrug NTM guideline-based antimycobacterial regimen at least 28 days prior to Screening due to lack of response or intolerance.
  Interventions: Drug: Molgramostim nebulizer solution; Device: PARI eFlow nebulizer system
- Group 3 (Experimental): Participants with chronic pulmonary MAC or MABSC infection not meeting recommendations for treatment with a multidrug NTM guideline-based antimycobacterial regimen based on failure to meet American Thoracic Society/Infectious Diseases Society of America (ATS/IDSA) criteria for NTM pulmonary disease (i.e. absence of radiologic findings and clinical symptoms beyond what is expected from underlying CF).
  Interventions: Drug: Molgramostim nebulizer solution; Device: PARI eFlow nebulizer system

INTERVENTIONS:
Drug: Molgramostim nebulizer solution — 300 µg / dose molgramostim (recombinant human GM-CSF) for inhalation
  Other Names: rhGM-CSF
Device: PARI eFlow nebulizer system — PARI eFlow nebulizer system

SUMMARY:
A study to evaluate the efficacy of inhaled molgramostim administered open-label to adult cystic fibrosis (CF) subjects with chronic pulmonary nontuberculous mycobacterial (NTM) infection, with or without ongoing antimycobacterial guideline based combination therapy.

DETAILED DESCRIPTION:
A Screening period will begin up to 10 weeks prior to the Baseline visit for collection of the sputum sample, but the remainder of the assessments including Safety labs will be completed within 6 weeks of Baseline, to determine eligibility. Adult participants with a history of CF and chronic pulmonary NTM infection will be considered for enrollment. Chronic pulmonary NTM infection will be defined by at least 3 positive NTM cultures (sputum or broncho-alveolar lavage (BAL)) for the same species/subspecies of mycobacterium avium (MAC) or mycobacterium abscessus complex (MABSC) within the 2 years prior to screening, with at least one positive within the past 6 months prior to screening and a minimum of 50% of NTM cultures positive over the past 2 years. Participants must additionally provide a positive sputum culture with the same species/subspecies obtained from the central laboratory during the Screening period to be eligible.

Three groups of participants will be recruited:

* Group 1: Participants with chronic pulmonary MAC or MABSC infection who have not consistently achieved negative NTM sputum cultures while currently on a multidrug NTM guideline-based antimycobacterial regimen, which has been ongoing for at least 9 months prior to the Baseline visit.
* Group 2: Participants with chronic pulmonary MAC or MABSC infection who remain sputum culture positive but have stopped a multidrug NTM guideline-based antimycobacterial regimen at least 28 days prior to Screening due to lack of response or intolerance.
* Group 3: Participants with chronic pulmonary MAC or MABSC infection not meeting recommendations for treatment with a multidrug NTM guideline-based antimycobacterial regimen based on failure to meet American Thoracic Society/Infectious Diseases Society of America (ATS/IDSA) criteria for NTM pulmonary disease (i.e. absence of radiologic findings and clinical symptoms beyond what is expected from underlying CF).

All participants will have Screening, Baseline, Week 1, 2 and followed by monthly Treatment visits from week 4 during the Treatment period. The Treatment period will be 48 weeks. Following the End of Treatment (Week 48), subjects will have a Follow-up visit at 4 and 12 weeks, and the End of Study visit 24 weeks after the End of Treatment. At the Baseline visit, eligible participants will start treatment with inhaled molgramostim.

At each visit any changes in concomitant medication will be recorded. Participants will be encouraged to contact the clinic between visits if they experience adverse events (AE), worsening of their condition or have any other concerns. If needed, unscheduled visits will be conducted at the Investigator's discretion. All participants will be maintained on their standard CF treatment and medications independent of NTM treatment status.

Treatment with inhaled molgramostim will be given at a dosage of 300 μg once daily for 48 weeks. Dosing will be done in the morning, after completion of the subject's normal airway clearance routine, where medications should be taken in the following order: bronchodilator, dornase alfa (Pulmozyme), inhaled antibiotics (e.g. TOBI) and lastly inhaled molgramostim.

Participants on a cyclical on-off anti-Pseudomonal regimen will have their trial visits (Baseline and subsequent visits in the Treatment Period) scheduled during a week after at least three weeks off treatment or after at least one week on-treatment of the antibiotic. Participants on a continuous inhaled regimen, including continuous alternating therapy (CAT), should have been on a stable regimen for at least 28 days prior to Baseline.

A data review will be conducted after the first 6 participants have completed 12 weeks of treatment. If safety concerns or poor tolerability are identified in this review, the review committee may decide on less frequent dosing for subsequent participants in the study. Additional safety reviews will be conducted at regular intervals thereafter. During the study, participants in Group 1 will continue use of antimycobacterial treatment, whereas participants in Groups 2 and 3 will receive inhaled molgramostim as monotherapy for their NTM infection. For participants in Group 1, the antimycobacterial therapy should preferably not change during the treatment period except in case of drug toxicity or adverse reactions. Antibiotics discontinued due to toxicity may be replaced, with drug selection and dose modification at the discretion of the treating physician. All changes in antimycobacterial treatment will be recorded, including reasons for each change. In the event the Investigator has evidence of infection while on treatment which requires more intensive therapy (i.e. additional antibiotics in Group 1 or addition of antibiotics to Group 2 or 3) the participant may be allowed to continue after discussion with the Sponsor medical monitor.

No formal sample size calculation was done as this is an initial pilot study. To be able to assess response in each of the three groups, a minimum of 8 participants with MAC or MABSC will be enrolled into each of the 3 groups, and a minimum of 30 participants will be enrolled across all 3 groups. The maximum number of participants enrolled into each group will be 12, and the maximum number of participants enrolled into the study will be 34.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from participant.
2. Confirmed diagnosis of CF according to the Cystic Fibrosis Foundation (CFF) 2017 Consensus Guidelines.
3. History of chronic pulmonary infection with M. avium complex (MAC) or M. abscessus complex (MABSC) (defined as at least three positive NTM cultures (sputum or BAL for the same species (MAC) or subspecies (MABSC) within the 2 years prior to the screening visit, with at least one positive within the past 6 months and a minimum of 50% of NTM cultures positive over the past 2 years) that does not demonstrate response to current treatment course based on decreasing NTM burden or frequency of positive cultures, and in the opinion of the Investigator is unlikely to resolve with current treatment course.
4. Subject fulfills criteria for inclusion in one of the following groups:

   Group 1: Subject with chronic pulmonary MAC or MABSC infection currently on a multidrug NTM guideline-based antimycobacterial regimen, which has been ongoing for at least 9 months prior to the Baseline visit.

   Group 2: Subject with chronic pulmonary MAC or MABSC infection who has stopped a multidrug NTM guideline-based antimycobacterial regimen at least 28 days prior to Screening due to lack of response or intolerance.

   Group 3: Subjects with chronic pulmonary MAC or MABSC infection not meeting recommendations for treatment with a multidrug NTM guideline-based antimycobacterial regimen based on failure to meet ATS/IDSA criteria for NTM pulmonary disease (i.e. absence of radiologic findings and clinical symptoms beyond what is expected from underlying CF).
5. Ability to produce sputum or be willing to undergo an induction protocol that produces sputum for clinical evaluation.
6. An additional sputum culture performed by the central laboratory, which is positive for the same species (MAC) or subspecies (MABSC) of NTM as before the trial within 10 weeks of Baseline.
7. CF which in the Investigator's opinion is clinically stable and not expected to require lung transplantation within the next year.
8. FEV1 ≥ 30% of predicted at screening that is normalized for age, gender, race, and height, using the Global Lung Function Initiative (GLI) equation.
9. Subjects who are co-infected with a respiratory pathogen, e.g. P. aeruginosa or S. aureus, must either be stable on a regular suppression antibiotic regimen or must be, in the opinion of the Investigator, stable despite the lack of such treatment.
10. Female or male ≥18 years of age.
11. If female, subjects who have been post-menopausal for more than 1 year or females of childbearing potential after a confirmed menstrual period using a highly efficient method of contraception (i.e. a method with less than 1% failure rate) during and until 30 days after last dose of trial treatment, having a negative serum pregnancy test at Screening (Visit 1) and a negative urine pregnancy test at dosing at Baseline (Visit 2) and must not be lactating.

    For purposes of this study, the Sponsor defines "acceptable methods of contraception" as:
    * Oral birth control pills administered for at least 1 monthly cycle prior to administration of the study drug.
    * A synthetic progestin implanted rod (eg, Implanon®) for at least 1 monthly cycle prior to the study drug administration but not beyond the 4th successive year following insertion.
    * Intrauterine devices (IUDs), inserted by a qualified clinician for at least 1 monthly cycle prior to study drug administration.
    * Medroxyprogesterone acetate (eg, Depo-Provera®) administered for a minimum of 1 monthly cycle prior to administration of the study drug and continuing through 1 month following study completion.
    * Hysterectomy or surgical sterilization.
    * Vasectomized partner
    * Abstinence.

    Double barrier method (diaphragm with spermicidal gel or condoms with contraceptive foam) is not considered an acceptable form of contraception.

    NOTE: For subjects prescribed Orkambi: Orkambi may substantially decrease hormonal contraceptive exposure, reducing the effectiveness and increasing the incidence of menstruation-associated adverse reactions. Hormonal contraceptives, including oral, injectable, transdermal, and implantable, should not be relied upon as an effective method of contraception when co-administered with Orkambi.
12. If male, subjects who, if sexually active of reproductive potential and non-sterile (i.e., male who has not been sterilized by vasectomy for at least 6 months and not diagnosed with infertility through demonstration of azoospermia in a semen sample and/or absence of vas deferens through ultrasound) are willing to use a barrier method of contraception, or their female partner must use an acceptable method of contraception, during the study and until 30 days after last dose of medication.
13. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures specified in the protocol as judged by the Investigator.

Exclusion criteria:

1. Use of non-maintenance antibiotic for a concurrent pulmonary or extrapulmonary infection within 28 days prior to the Baseline visit.
2. Use of a maintenance antibiotic regimen containing azithromycin for a concurrent non-NTM pulmonary infection within 28 days prior to the Baseline visit. For subjects in Group 1, azithromycin is allowed if part of ongoing multidrug NTM guideline-based antimycobacterial regimen.
3. Prior therapy with inhaled or systemic granulocyte macrophage colony stimulating factor (GM-CSF).
4. Subjects with hemoptysis of ≥60 mL in a 24-hour period within 4 weeks prior to Screening.
5. Life expectancy of less than 6 months according to Investigator's judgement.
6. History of, or present, myeloproliferative disease, leukemia or other hematological malignancy.
7. Active pulmonary malignancy (primary or metastatic); or any malignancy requiring chemotherapy or radiation therapy within 1 year prior to Screening or anticipated during the study period.
8. Active autoimmune disorder or other condition requiring therapy associated with significant immunosuppression, e.g. such as systemic corticosteroids at a dose equivalent of 10 mg/day or more of prednisolone or other significant immunosuppressant medications, within 3 months prior to Screening or anticipated during the study period. Inhaled or topical corticosteroids, or brief courses (<14 days) of systemic corticosteroids for pulmonary exacerbations or other self-limited conditions are permitted.
9. Changes in antimicrobial, bronchodilator, anti-inflammatory or corticosteroid medications, or changes in Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) modulators, within 28 days prior to the Baseline visit.
10. Pulmonary tuberculosis requiring treatment or treated within 2 years prior to Screening.
11. History of human immunodeficiency virus (HIV) infection or other disease associated with significant immunodeficiency.
12. History of lung or other solid organ transplantation or currently on the list to receive lung or other solid organ transplantation.
13. History of congestive heart failure (CHF) New York Heart Association (NYHA) Class III or greater in severity.
14. History of cardiovascular ischemic event within 6 months of Baseline.
15. Any change in chronic NTM multi-drug antimycobacterial regimen within 28 days prior to Screening.
16. Treatment with any investigational medicinal product within 28 days of Screening.
17. Previous experience of severe and unexplained side-effects during aerosol delivery of any kind of medicinal product.
18. Any other condition that, in the opinion of the Investigator, would preclude informed consent or assent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Nick, MD, Principal Investigator — National Jewish Health
Locations (5):
- United States (5):
  - National Jewish Health, Denver, Colorado
  - Central Florida Pulmonary Group, Orlando, Florida
  - Northwell Health, New Hyde Park, New York
  - University of North Carolina at Chapel Hill - UNC Marisco Clinical Research Center, Chapel Hill, North Carolina
  - UT Southwestern Medical Center Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 sites in US participated in the study. The first participant was enrolled on 20 June 2019 and last participant completed the study on 2 October 2020, the same date the study was terminated.
Pre-assignment Details: A total of 28 subjects were screened for the trial. Fourteen subjects were screening failures.
Groups:
- Not Consistently NTM Sputum Negative: Participants with chronic pulmonary MAC or MABSC infection who have not consistently achieved negative NTM sputum cultures while currently on a multidrug NTM guideline-based antimycobacterial regimen, which has been ongoing for at least 9 months prior to the Baseline visit.
  Molgramostim nebulizer solution: 300 µg / dose molgramostim (recombinant human GM-CSF) for inhalation
  PARI eFlow nebulizer system: PARI eFlow nebulizer system
- NTM Sputum Positive: Participants with chronic pulmonary MAC or MABSC infection who remain sputum culture positive but have stopped a multidrug NTM guideline-based antimycobacterial regimen at least 28 days prior to Screening due to lack of response or intolerance.
  Molgramostim nebulizer solution: 300 µg / dose molgramostim (recombinant human GM-CSF) for inhalation
  PARI eFlow nebulizer system: PARI eFlow nebulizer system
- Did Not Meet Recommendations for Treatment With a Multidrug NTM Antimycobacterial Treatment: Participants with chronic pulmonary MAC or MABSC infection not meeting recommendations for treatment with a multidrug NTM guideline-based antimycobacterial regimen based on failure to meet American Thoracic Society/Infectious Diseases Society of America (ATS/IDSA) criteria for NTM pulmonary disease (i.e. absence of radiologic findings and clinical symptoms beyond what is expected from underlying CF).
  Molgramostim nebulizer solution: 300 µg / dose molgramostim (recombinant human GM-CSF) for inhalation
  PARI eFlow nebulizer system: PARI eFlow nebulizer system
Period: Overall Study
Arm/Group | Not Consistently NTM Sputum Negative | NTM Sputum Positive | Did Not Meet Recommendations for Treatment With a Multidrug NTM Antimycobacterial Treatment
Started | 7 | 3 | 4
Completed | 0 | 0 | 0
Not Completed | 7 | 3 | 4
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Withdrawal due to Covid-19 | 3 | 0 | 0
Not completed — Sponsor decision to terminate study | 3 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 7 | 3 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (11.78) | 46.3 (20.03) | 38.8 (12.28) | 35.5 (14.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 7
  Male | 4 | 1 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 7 | 3 | 3 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Causative species/ subspecies [Count of Participants; unit: Participants]
  Mycobacterium abscessus ss abscessus | 6 | 3 | 1 | 10
  Mycobacterium abscessus ss massiliense | 1 | 0 | 0 | 1
  Mycobacterium avium | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sputum NTM Culture Conversion to Negative
Description: NTM sputum culture conversion to negative (defined as at least three consecutive negative mycobacterial cultures collected at least 4 weeks apart during the treatment period).
Time Frame: 48 weeks
Population: Safety analysis set (participants who received at least one dose of trial treatment).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 7 | 3 | 4
Participants | 3 | 1 | 3

2. Secondary Outcome: Number of Participants With NTM Sputum Culture Microbiological Cure
Description: NTM sputum culture microbiological cure (defined as multiple consecutive negative but no positive cultures with the causative species after last culture conversion and until the end of treatment (Week 48)).
Time Frame: 48 weeks
Population: Safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 7 | 3 | 4
Participants | 1 | 1 | 1

3. Secondary Outcome: Time to First NTM Sputum Culture Conversion
Description: Time to first NTM sputum culture conversion during the treatment period.
Time Frame: 48 Weeks
Population: Only participants who had NTM sputum culture conversion during the treatment period were analyzed. The mean survival time and its standard error of the mean were underestimated because the largest observation was censored and the estimation was restricted to the largest event time.
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 3 | 1 | 3
weeks | 23.21 (1.991) | 8.57 | 21.54 (1.933)

4. Secondary Outcome: Number of Participants With Sputum Smear Conversion to Negative
Description: Sputum smear conversion to negative (defined as at least three consecutive negative acid-fast bacilli stained sputum smears on microscopy, collected at least 4 weeks apart in subjects who were smear positive at baseline) during the treatment period.
Time Frame: 48 weeks
Population: Safety analysis set. Only participants who had positive smear at baseline were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 2 | 0 | 0
Participants | 2 | 0 | 0

5. Secondary Outcome: Number of Participants With Consistent Sputum Smear Conversion to Negative Treatment (Week 48) in Subjects Who Were Smear Positive at Baseline)
Description: Consistent sputum smear conversion to negative (defined as multiple consecutive negative but no positive smears after last smear conversion and until the end of treatment (Week 48) in subjects who were smear positive at baseline).
Time Frame: 48 weeks
Population: Safety analysis set. Only participants who had positive smear at baseline were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 2 | 0 | 0
Participants | 1 | 0 | 0

6. Secondary Outcome: Time to First NTM Sputum Smear Conversion
Description: Time to first NTM sputum smear conversion during the treatment period.
Time Frame: 48 weeks
Population: Safety analysis set. Only participants who had positive smear at baseline were analyzed. The mean survival time and its standard error were underestimated because the largest observation was censored and the estimation was restricted to the largest event time.
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 2 | 0 | 0
weeks | 14.55 (2.084) |  |

7. Secondary Outcome: Number of Participants With Durable NTM Sputum Microbiological Cure
Description: Durable NTM sputum microbiological cure for the NTM isolate(s) treated without recurrence at Week 12 after end of treatment.
Time Frame: 12 weeks after end of treatment
Population: Safety analysis set. Only participants who had positive smear at baseline were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 2 | 0 | 0
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs) were assessed on or after the first dose of trial drug to 28 days after last dose.
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/7 | 1/3 | 1/4
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=7) | Group 2 (N=3) | Group 3 (N=4)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=7) | Group 2 (N=3) | Group 3 (N=4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 2 | 2
Fatigue (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Complication associated with device (General disorders) | 1 | 0 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 1 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Localised infection (General disorders) | 0 | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 2 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 1
Albumin urine present (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood chloride decreased (Investigations) | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0
Glucose urine present (Investigations) | 1 | 0 | 0
Specific gravity urine decreased (Investigations) | 1 | 0 | 0
Urine ketone body present (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Parotid duct obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Insomina (Psychiatric disorders) | 1 | 0 | 0
Mania (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, some specified endpoints had insufficient data to be analyzed:

* Durable NTM sputum smear conversion to negative without subsequent positive smears at Week 12 after End of Treatment (EOT).

Change from Baseline to EOT and Week 12 after EOT in:

* semi-quantitative grade of number of NTM on microscopy of AFB stained sputum smears
* FEV1 (percent predicted)
* respiratory domain score assessed by CFQ-R
* body mass index

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT03597347/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT03597347/SAP_001.pdf